CLINICAL TRIAL: NCT00073138
Title: A Phase 2 Study of ABT-751 in Subjects With Refractory Colorectal Carcinoma
Brief Title: A Study of ABT-751 in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-446
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ABT751

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-751

SUMMARY:
The purpose of the study is to determine if ABT-751 will decrease tumors, and determine how long the tumor shrinkage can be maintained in patients with colorectal cancer. Patients will receive ABT-751 by mouth daily for 21 days. Patients will be off drug for 7 days before starting the next cycle of drug.

ELIGIBILITY:
Inclusion Criteria

* Colorectal cancer.
* Recurrent tumor following treatment with irinotecan and/or oxaliplatin.
* Able to tolerate normal activities of daily living.
* Adequate bone marrow, kidney, and liver function.

Exclusion Criteria

* Pregnant or breast feeding.
* Anti-tumor therapy within 4 weeks of the start of ABT-751 administration.
* Prior radiation therapy.
* CNS metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate in subjects with Recurrent Colorectal Cancer | 1 year

SECONDARY OUTCOMES:
Time to Tumor Progression (TTP) | 1 year
Survival | 2 years
Toxicities associated with treatment administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Eliopoulos, MD, Study Director — Abbott
Locations (6):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin Medical Center, Madison, Wisconsin